CLINICAL TRIAL: NCT04975347
Title: Opioid Antagonism in Individuals Ascertained Through the Partners HealthCare Biobank
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stephanie B. Seminara, MD (Other)
Responsible Party: Sponsor-Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 313512
Record Dates: First submitted 2021-07-15; First posted 2021-07-23 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Reproductive Disorders
Keywords: naloxone
MeSH Terms: interventions — Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (No Intervention): one period of frequent blood sampling with no medication administered
- Arm 2 (Experimental): one period of frequent blood sampling with no medication administered; one period of frequent blood sampling with IV administration of naloxone (one bolus and an infusion over an up to 12-hour period.)
  Interventions: Drug: Naloxone

INTERVENTIONS:
Drug: Naloxone — One bolus and one infusion of naloxone
  Arms: Arm 2

SUMMARY:
The goal of this study is to evaluate the effects of opioid antagonists on the hypothalamic-pituitary-gonadal axis in healthy subjects.

DETAILED DESCRIPTION:
Arm 1 Assignment: Individuals will be assigned to group 1 or group 2 based on their genetic features.

Arm 2 Assignment: Each study subject will serve as their own control.

Delivery of Interventions:

* Prior to the study visit, subjects will undergo a review of their medical history and screening laboratories.
* During the study, the subjects will complete the following

  * Arm 1: Undergo frequent blood sampling for up to 12 hours
  * Arm 2:

    * Period 1: Blood sampling q10 min for up to 12 hours
    * Period 2: Blood sampling q10 min for up to 12 hours with concurrent administration of naloxone bolus followed by a naloxone infusion

ELIGIBILITY:
Inclusion

* Age 18-45 years (women) OR 18-60 years (men)
* Genetic sequencing data available via Mass General Brigham Biobank
* All medical conditions stable and well controlled
* If applicable, willing to use birth control methods (as approved by a study medical professional) during protocol participation
* Normal blood pressure (systolic BP < 140 mm Hg, diastolic < 90 mm Hg)
* Negative urine drug screening panel
* Hemoglobin within sex-specific reference range
* For women, negative serum hCG pregnancy test

Exclusion

* Any condition (medical, mental, or behavioral) that, in the opinion of a study investigator, would likely interfere with participation in/completion of the protocol
* Current or recent use of a medication (including hormonal replacement) that, in the opinion of a study investigator, can modulate the reproductive axis and, if applicable, unwilling to complete an appropriate washout for that particular medication and its method of administration
* Current or recent use of a medication that affects the opioid pathway
* Active illicit drug use
* Excessive alcohol consumption (> 10 drinks/week)
* For women, pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Average change in Luteinizing Hormone (LH) pulse frequency | Two 12-hour periods
  Change in LH pulse frequency before and during naloxone infusion
Difference in Average LH Pulse Frequency | one 12-hour period
  difference in LH pulse frequency between variant-carriers and control participants

SECONDARY OUTCOMES:
Average change in LH pulse amplitude | Two 12-hour periods
  Change in LH pulse amplitude before and during naloxone infusion

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No